CLINICAL TRIAL: NCT04007692
Title: Suturing Pattern for Endolumenal Stenting Procedures
Brief Title: Optimal Endoscopic Suturing Pattern for Esophageal Stent Fixation
Status: Terminated | Type: Observational
Why Stopped: Accrual difficulties:
  This trial was initiated prior to COVID-19 and interrupted by the pandemic for a significant length of time.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Barham K. Abu Dayyeh, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 18-003817
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Stenosis; Stent Migration; Suture, Complication
Keywords: Esophageal stenosis; Endoscopic suturing; Esophageal stent fixation; Stent migration
MeSH Terms: conditions — Esophageal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Simple interrupted suture group: Participants will have a simple interrupted suturing pattern, determined by care provider, at the time of esophageal stent placement for esophageal stent fixation as part of standard care and will have an endoscopy at 3-4 weeks after the stent placement as part of a routine follow-up.
  Interventions: Procedure: Esophageal stent placement
- Triangular suture group: Participants will have a triangular suturing pattern, determined by care provider, at the time of esophageal stent placement for esophageal stent fixation as part of standard care and will have an endoscopy at 3-4 weeks after the stent placement as part of a routine follow-up.
  Interventions: Procedure: Esophageal stent placement

INTERVENTIONS:
Procedure: Esophageal stent placement — Exposure of interest is standard of care esophageal stent placement

SUMMARY:
Researchers are trying to determine which suturing pattern for esophageal stent placement is more effective in a randomized fashion as currently what suturing pattern to use is an arbitrary decision.

DETAILED DESCRIPTION:
The participants who are receiving esophageal stent placement will be prospectively randomized to receive two suturing patterns (simple interrupted pattern and triangular pattern) for endoscopic esophageal stent fixation. We will investigate rate of the stent migration at 3-4 weeks by endoscopy after the stent placement as part of routine clinical care. Data of the duration of endoscopic suturing, adverse events, details of the stent used, indication for use will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 or above
* Subjects undergoing esophageal stent placement with any indication

Exclusion Criteria:

* Imprisoned individuals,
* Institutionalized patients
* Inability or unwillingness of individual

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-vulnerable adults who are receiving an endoscopically placed esophageal stent for any indication at Mayo Clinic Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Stent migration rate | 4 weeks post stent placement
  Number of participants with stent migration as assessed by objective evidence of stent migration on endoscopy at 3-4 weeks after esophageal stent placement
Adverse Events | 4 weeks
  Number of adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Barham K Abu Dayyeh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials